CLINICAL TRIAL: NCT04810299
Title: Evaluation of the Effect of Aromatherapy Massage Applied to Patients After Colorectal Surgery on Early Symptom Control
Brief Title: Effect of Aromatherapy Massage on Symptom Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Özge Yaman, Principal İnvestigator, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Özge YAMAN
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
Keywords: aromatherapy; foot massage; anxiety; pain; sleep quality; fatigue
MeSH Terms: conditions — Colorectal Neoplasms; Anxiety Disorders; Pain; Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aromatherapy Massage Group (Experimental): According to this Tisserand Institute guide chart, for a 2% dilution process, dilution will be provided with a total of 12 drops by adding 4:4:4 drops of lavender, Roman chamomile and ginger essential oils in 20 ml of sweet almond oil. Expert opinion was obtained from a phytotherapy and aromatherapy specialist physician that the oils and dilution rates used were appropriate. Foot massage will be applied on the 1st, 2nd and 3rd postoperative days. State Anxiety Scale, Visual Analogue Scale (VAS-F), Visual Analogue Scale (VAS-P), Post-operative Nausea-Vomiting Impact Scale will be applied before and after the application.Richard-Campbell Sleep Quality Scale will be applied before application Foot massage will be applied for 20 minutes.
  Interventions: Other: Aromatherapy
- Classical Foot Massage Group (Experimental): Baby oil will be applied as massage oil to patients who are assigned to the classical foot massage group before the surgery. Foot massage will be applied for 20 minutes on the 1st,2nd and 3rd days. State Anxiety Scale, Visual Analogue Scale (VAS-F), Visual Analogue Scale (VAS-P), Post-operative Nausea-Vomiting Impact Scale will be applied before and after the application.Richard-Campbell Sleep Quality Scale will be applied before application
  Interventions: Other: Classical foot massage
- Control Group (No Intervention): Except for routine care practices, no attempt will be made to the patients assigned to the pre-operative control group. State Anxiety Scale, Richard-Campbell Sleep Quality Scale, Visual Analogue Scale (VAS-F), Visual Analogue Scale (VAS-P), Post-operative Nausea-Vomiting Impact Scale will be applied on postoperative 1st, 2nd and 3rd days. The same scales will be re-evaluated 60 minutes after the first measurement. Richard-Campbell Sleep Quality Scale will be applied once

INTERVENTIONS:
Other: Aromatherapy — Aromatherapy; It is one of the complementary therapy methods defined as the therapeutic use of essential oils obtained from parts of plants such as root, seed, leaf, flower, shell with appropriate methods.
  Arms: Aromatherapy Massage Group
Other: Classical foot massage — Classical foot massage; It is defined as a massage technique based on the principle of systematic relaxation
  Arms: Classical Foot Massage Group

SUMMARY:
Although the incidence of colorectal cancers is high, it is often possible to treat it when diagnosed at an early stage. Although the treatment options vary according to many factors such as the type and stage of the cancer, possible side effects, the preference of the patient, and the general health status, surgery stands out as the most commonly used treatment method. However, in addition to the methods and drugs used in the diagnosis and treatment process, temporary or permanent stomas that are opened to ensure discharge cause biopsychosocial effects on the life of the individual and lead to deterioration of the quality of life. In this context, knowing and resolving the problems experienced by patients in the pre-operative and post-surgical period, which is the most commonly used treatment method, will also increase the quality of life of patients. In the literature, it was stated that patients experienced high levels of anxiety before colorectal surgery and this situation caused emotional and cognitive reactions; in the postoperative period, it is seen that they experience many problems such as anxiety, restlessness, fatigue, gastrointestinal dysfunction, pain, loss of control (inability to control gas and stool output), decreased appetite, insomnia, nausea-vomiting, abdominal distension, constipation. However, modern treatment methods, drug and non-drug treatments used to control these symptoms are not effective in some cases. At this stage, complementary and alternative medicine applications come into play, one or more of these methods are used to alleviate symptoms and increase well-being during traditional treatments. In this study, it was planned to evaluate the effect of aromatherapy massage after colorectal surgery on postoperative symptom control (pain, anxiety, fatigue, sleep quality, nausea-vomiting, flatulence).

DETAILED DESCRIPTION:
The population of the study will consist of patients who underwent colorectal cancer surgery between June 2021 and June 2022, and the sample of patients who meet the criteria for inclusion in the study.The sample was planned to be 90 people, 30 patients for each of the aromatherapy massage, classical foot massage and control groups. However, power analysis was also performed to calculate the minimum sample size to be reached. In the study, it was aimed to evaluate the differences in mean scale between three groups, including one control and two experiments. When it is not known how many units of difference between groups are important, the effect width value is taken as 0.35 as the method used. The effect width value gives results with a very high constraint of 0.10, medium level of 0.25 and a maximum acceptance constraint of 0.40. The total number of patients was 84, including 28 patients in the groups, with an error margin of 5% and a width of effect value of 0.35 at 81.19% power level.Block Randomization technique will be used in the sample selection of the research. In order to blind the randomization, it was made by a statistician who was not related to the research and the group rankings were put in 9 envelopes and numbered by another person who was not related to the research. For data collection Patient Information Form , Visual Analog Scale (VAS-Pain), Visual Analog Scale (VAS-Fatigue), Richard-Campbell Sleep Quality Scale, State Anxiety Scale, Post-operative Nausea-Vomiting Effect Scale will be used.The first interview with the patients will be held in the preoperative period and information will be given about the research. For patients who agree to participate in the study, a Patient Information Form will be filled out and a group assignment will be made using the block randomization method.

ELIGIBILITY:
Inclusion Criteria:

* Are over the age of 18
* Can understand and speak Turkish
* No mental or neurological disorders that may affect communication skills
* Not allergic to aromatic oils for aromatherapy massage group
* Patients undergoing curative surgery
* Not using antidepressant medication
* With an ASA score of 1-2-3
* Undergoing elective surgery
* Follow-up in the service after surgery
* No secondary cancer and recurrence surgery
* No contraindications for foot massage
* No major complications (bleeding, obstruction, anastomotic leak etc.) during the postoperative period
* Individuals who agree to participate in the study will be included.

Exclusion Criteria:

* Under the age of 18
* Cannot understand and speak Turkish
* Having a mental or neurological condition that affects communication skills
* For aromatherapy massage group, allergic to aromatic oils
* Having had aromatherapy practice before
* Refusing to participate in research
* Stage IV patients
* Using antidepressant medication
* Emergency surgery applied
* ASA score of 4-5
* Permanent stoma opening
* Follow-up in intensive care after surgery
* Secondary cancer or surgery after relapse
* Major complications during the postoperative period
* Contraindicated for foot massage application (paraplegia, acute gout, foot ulcer, thrombosis, peripheral vascular disease, diffuse edema or lymphedema, acute foot injury or fracture)
* Having a pacemaker, uncontrolled hypertension, uncontrolled thyroid problems, epilepsy, bladder or kidney stones
* Patients with signs of active infection and fever will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Pain levels | The change between the first, second and third days after surgery will be checked.
  A visual analog scale will be used, with a score expressing painlessness on one side and unbearable pain on the other. Their values range from 0-10. Absence of pain is defined as "0 points" and unbearable pain is defined as "10 points".
Anxiety levels | The change between the first, second and third days after surgery will be checked.
  Measurements will be made using the State Anxiety Scale. This scale determines how the individual feels at a particular moment and under certain conditions.
Fatigue levels | The change between the first, second and third days after surgery will be checked.
  A visual analog scale will be used.Their values range from 0-10.
Sleep quality | The change between the first, second and third days after surgery will be checked.
  The Richard-Campbell Sleep Quality Scale will be used. This scale evaluates the depth of night sleep, the duration of falling asleep, the frequency of awakening, the duration of being awake when awakened, the quality of sleep, and the noise level in the environment.
Nausea-vomiting | The change between the first, second and third days after surgery will be checked.
  There are four options in the Post-operative Nausea Vomiting Impact Scale, which consists of two questions, with 0, 1, 2, 3 points for each question. The first question is whether there is vomiting or retching, the frequency is questioned, the second question is whether there is nausea (feeling of discomfort in the stomach and vomiting), if there is a feeling of nausea, you can get out of bed, move comfortably in bed, walk normally or your daily life activities such as eating and drinking. whether it affects or not is questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek AYGİN, PhD, Study Director — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is planned to be published after the study is completed.

REFERENCES:
- [Derived] Yaman O, Aygin D, Altintoprak F, Guclu E. The effects of aromatherapy massage given to patients after colorectal cancer surgery on symptom management: A randomized controlled study. Complement Ther Clin Pract. 2024 Nov;57:101900. doi: 10.1016/j.ctcp.2024.101900. Epub 2024 Sep 2. PMID 39241341